CLINICAL TRIAL: NCT05111236
Title: Potential Benefits of Home Based Exercise Programs With and Without Traditional Massage in the Management of Spastic Cerebral Palsy: A Randomized Controlled Trial.
Brief Title: Potential Benefits of Home Based Exercise Programs in the Management of Spastic Cerebral Palsy
Acronym: HEP&CP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Rehabilitation Medicine, Islamabad, Pakistan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIRM-Physio/01
Record Dates: First submitted 2021-10-28; First posted 2021-11-08 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-10

CONDITIONS: Cerebral Palsy, Spastic, Diplegic
Keywords: cerebral palsy, massage, spasticity, motor function
MeSH Terms: conditions — Cerebral palsy, spastic, diplegic; Cerebral Palsy; Muscle Spasticity | interventions — Medicine, Thai Traditional

STUDY DESIGN:
Intervention Model Description: It is a RCT with two groups, RPT and Massage. Both groups will receive routine physical therapy (with addition of traditional massage in Massage group only) five days a week for a period of 12 weeks.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be kept blind about group allocation and identification of the participants before assessments at baseline, after 06 weeks and 12 weeks of intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RPT Group (Active Comparator): Routine physical therapy comprising stretching of spastic muscles, Strengthening of weak muscles, positioning ( how to make sitting and standing postures at home) and posturing strategies. This whole regimen will be practiced fives times a week for a period of twelve weeks.
  Other Names:
  • Routine Physical Therapy
  Interventions: Other: Routine physical therapy
- Massage Group (Experimental): Traditional massage of thirty minutes duration ( five minutes of massage will be provided to all four limbs, front and back of trunk area) prior to routine physical therapy. Routine physical therapy comprising stretching of spastic muscles, Strengthening of weak muscles, positioning ( how to make sitting and standing postures at home) and posturing strategies.
  Other Names:
  • Routine physical therapy and Traditional massage
  Interventions: Other: Routine physical therapy; Other: Traditional massage

INTERVENTIONS:
Other: Routine physical therapy — Rehabilitation strategies in management of children with spastic CP
Other: Traditional massage — Rehabilitation strategies in management of children with spastic CP
  Arms: Massage Group

SUMMARY:
The study will be conducted to see the potential benefits of home based exercise program comprising routine physical therapy and traditional massage in the management of spastic cerebral palsy (CP). It will be a randomized controlled trial having two groups, RPT group and Massage group. Both groups will be provided with routine physical therapy treatment comprising stretching of spastic muscles, strengthening of weak muscles, positioning and posturing strategies. Massage group will also receive traditional massage in addition to routine physical therapy. Parents/Caregivers will be trained to perform routine physical therapy and traditional massage at home. Data will collected using a structured questionnaire, Modified Ashworth Scale (MAS), Gross Motor Function Measure (GMFM),Gross Motor Function Classification System (GMFCS) and CP Child's Caregiver Priorities & Child Health Index of Life with Disabilities at baseline, after 6th and 12th weeks of intervention.

DETAILED DESCRIPTION:
CP is among the most common type of physical disabilities presenting itself in children across the globe. Although its incidence range has been reported from 2 to 2.5 cases per 1000 live births globally, however it may be many folds in poor counties due to lack of reporting and absence of CP registries at national level . Many interventions are in use to manage the disabling and lifelong consequences of this condition. However majority of these interventions remain beyond the reach of poor population especially in under developed countries with poor socio-economic status like Pakistan. This creates a need for search to such interventions which should be locally available, accessible, low cost, affordable, and doable by the poor population so that disabling consequences of this condition may be minimized. RPT and traditional massage performed by parents at home after proper training fall in the category of such low cost interventions. Hence there is dire need to investigate the potential benefits of such interventions. That is why this RCT has been planned.

ELIGIBILITY:
Inclusion Criteria:

* Child should have established diagnosis of spastic cerebral palsy (diplegic types only).

Exclusion Criteria:

* Children having moderate to severe contractures.

  * Children having moderate to severe mental retardation and with multiple disabilities.
  * Children with Attention Deficit Hyperactive Disorder (ADHD), uncontrolled seizures and behavioral disorders

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth scale (MAS) | Twelve weeks
  0 = No increase in muscle tone
  * 1 = Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  * 1+ = Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the Range Of Motion (ROM)
  * 2 = More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  * 3 = Considerable increase in muscle tone, passive movement difficult.
  * 4 = Affected part(s) rigid in flexion or extension

SECONDARY OUTCOMES:
Gross motor Function Measure (GMFM-88) | Twelve weeks
  It is used to check the gross motor ability having total of 88 items to be checked in 05 different domain Lying and Rolling (total score 51), Sitting (Total score 60), Crawling and Kneeling( total 42), standing (total 39), walking running jumping (total 72)
Gross Motor Function Classification System (GMFCS) | Twelve weeks
  It has five levels I to V showing the mobility level. Level I to III represent ambulatory status while IV and V represent Non- ambulatory status
CPCHILD ( Caregiver Priorities & child health index of life with Disabilities | Twelve weeks
  It is used to check the quality of life of children with cerebral palsy. It has 09 sections to be completed representing different states related to quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Qamar Mahmood, Principal Investigator — HOD, Physiotherapy Department
Locations (1):
- National Institute of Rehabilitation Medicine (NIRM), Islamabad, Federal Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirby RS, Wingate MS, Van Naarden Braun K, Doernberg NS, Arneson CL, Benedict RE, Mulvihill B, Durkin MS, Fitzgerald RT, Maenner MJ, Patz JA, Yeargin-Allsopp M. Prevalence and functioning of children with cerebral palsy in four areas of the United States in 2006: a report from the Autism and Developmental Disabilities Monitoring Network. Res Dev Disabil. 2011 Mar-Apr;32(2):462-9. doi: 10.1016/j.ridd.2010.12.042. Epub 2011 Jan 26. PMID 21273041
- [Background] Reddihough DS, Collins KJ. The epidemiology and causes of cerebral palsy. Aust J Physiother. 2003;49(1):7-12. doi: 10.1016/s0004-9514(14)60183-5. PMID 12600249
- [Background] Bhasin TK, Brocksen S, Avchen RN, Van Naarden Braun K. Prevalence of four developmental disabilities among children aged 8 years--Metropolitan Atlanta Developmental Disabilities Surveillance Program, 1996 and 2000. MMWR Surveill Summ. 2006 Jan 27;55(1):1-9. PMID 16437058
- [Background] Reddihough DS, Jiang B, Lanigan A, Reid SM, Walstab JE, Davis E. Social outcomes of young adults with cerebral palsy. J Intellect Dev Disabil. 2013 Sep;38(3):215-22. doi: 10.3109/13668250.2013.788690. Epub 2013 May 14. PMID 23672634
- [Background] Hurvitz EA, Leonard C, Ayyangar R, Nelson VS. Complementary and alternative medicine use in families of children with cerebral palsy. Dev Med Child Neurol. 2003 Jun;45(6):364-70. doi: 10.1017/s0012162203000707. PMID 12785436
- [Background] Novak I, McIntyre S, Morgan C, Campbell L, Dark L, Morton N, Stumbles E, Wilson SA, Goldsmith S. A systematic review of interventions for children with cerebral palsy: state of the evidence. Dev Med Child Neurol. 2013 Oct;55(10):885-910. doi: 10.1111/dmcn.12246. Epub 2013 Aug 21. PMID 23962350
- [Background] Mahmood Q, Habibullah S, Babur MN. Potential effects of traditional massage on spasticity and gross motor function in children with spastic cerebral palsy: A randomized controlled trial. Pak J Med Sci. 2019 Sep-Oct;35(5):1210-1215. doi: 10.12669/pjms.35.5.478. PMID 31488980
- [Background] Novak I, Berry J. Home program intervention effectiveness evidence. Phys Occup Ther Pediatr. 2014 Nov;34(4):384-9. doi: 10.3109/01942638.2014.964020. Epub 2014 Oct 15. No abstract available. PMID 25317927
- [Derived] Mahmood Q, Habibullah S, Aurakzai HU. Effectiveness of simple and basic home-based exercise programs including pediatric massage executed by caregivers at their homes in the management of children with spastic cerebral palsy: A randomized controlled trial. J Pediatr Rehabil Med. 2024;17(1):97-106. doi: 10.3233/PRM-220135. PMID 38427509